CLINICAL TRIAL: NCT01783717
Title: Effects of Exenatide on Obesity and/or Diabetes Mellitus Due to Hypothalamic Damage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, Clinical Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-217
Record Dates: First submitted 2012-12-25; First posted 2013-02-05 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Hypothalamic Obesity; Diabetes Mellitus
MeSH Terms: conditions — Sexual Infantilism; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exenatide (Experimental): 5mcg twice a day for 4 weeks increased to 10 mcg twice a day for 8 weeks
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — 5mcg twice a day for 4 weeks increased to 10 mcg twice a day for 8 weeks
  Other Names: Byetta

SUMMARY:
The purpose of this study is to examine the effect of exenatide on body weight and glycemic control in subjects with obesity and/or diabetes mellitus due to hypothalamic damage.

DETAILED DESCRIPTION:
Patients with hypothalamus lesion caused by tumors in the hypothalamic region, such as craniopharyngioma and germ cell tumors, and inflammatory diseases are susceptible to develop severe obesity and diabetes mellitus. The occurrence of hypothalamic obesity in patients after surgery with or without radiotherapy for craniopharyngioma can be as high as 42-66%, and the incidence of type 2 diabetes mellitus of them is twice as much as healthy controls. Treatment of obesity and diabetes mellitus in this population is crucial for increasing morbidity and mortality. However, diet and exercise intervention has been proven useless in previous studies. Safe and effective medicine remains to be developed. Exenatide, a GLP-1 receptor agonist, which play an antihyperglycemic role through a variety of mechanisms, such as enhancing glucose-dependent insulin secretion, increasing beta cell mass and decreasing glucagon secretion, possesses a potent ability to induce satiety, slow gastric emptying and reduce food intake, resulting in weight loss both in diabetics and patients with simple obesity. Previous animal study has already shown GLP-1 agonist exendin-4 leads to reduction of weight and caloric intake in a rat model of hypothalamic obesity. Therefore, the investigators hypothesize exenatide treatment might lead to weight loss in hypothalamic obese patients and improve their glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 55 years old;
2. Greater than 6 months post-treatment (including surgery, radiotherapy or chemotherapy) of craniopharyngioma or other diseases in the hypothalamic region;
3. BMI≧28kg/m2 and/or diabetes mellitus;
4. Greater than 3 months after adequate replacement therapy for hypothalamic-pituitary-adrenal (HPA) axis and hypothalamic-pituitary-thyroid (HPT) axis;
5. Sign informed consent document.

Exclusion Criteria:

1. Less than 6 months post surgery or radiotherapy or chemotherapy for craniopharyngioma or other diseases in the hypothalamic region;
2. Inadequate replacement for the HPA axis and HPT axis or undertaking adjustments of the kind or dose of the substitutive medicine;
3. Use of weight loss drugs or initiation of a weight loss program within past 3 months;
4. Use of GLP-1 agonists or analogues or dipeptidyl peptidase IV (DPP-IV) inhibitors within past 3 months;
5. History of bariatric surgery;
6. Diagnosed with simple obesity or diabetes mellitus prior to the hypothalamic disorders, and those diagnosed with type 1 diabetes mellitus;
7. With end-stage-renal diseases or history of kidney transplant or complicated with acute/chronic kidney failure (GFR≦30ml/min);
8. History of inflammatory bowel diseases or gastroparesis or other gastric mortility problems;
9. History of pancreatitis or chronic cholecystitis;
10. History of allergic reaction to exenatide or other medication components;
11. Undertaking warfarin;
12. Pregnant or lactating women;
13. Are participating in, or have participated in other drug clinical trials within past 3 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-01 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change in body weight frome baseline to end of the study. | 3 months
BMI | baseline and 3 months
HbA1c | baseline and 3 months
Blood glucose level. | 3 months.
Beta cell function. | baseline and 3 months
Insulin sensitivity. | baseline and 3 months

SECONDARY OUTCOMES:
Waistline | baseline and 3 months
Ratio of body fat | baseline and 3 months
The amount of daily energy intake | baseline and 3 months
Resting energy expenditure (kcals per day) | baseline and 3 months
Grade of metabolic equivalents (MET) scales | baseline and 3 months
Hipline. | baseline and 3 months
waistline/hipline ratio | baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Li yi ming, Principal Investigator — Huashan Hospital
Locations (1):
- Department of Endocrinology and Metabolism, Shanghai, Shanghai Municipality, China